CLINICAL TRIAL: NCT03028272
Title: Hearing Results and Post Surgical Outcomes Using Amniotic Membrane Allograft Versus Fascia for Tympanoplasty: A Randomized Prospective Trial
Brief Title: Hearing Results and Post Surgical Outcomes Using Amniotic Membrane Allograft vs. Fascia for Tympanoplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of qualified participants
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Arnaldo L. Rivera, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006074
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Tympanic Membrane Perforation
Keywords: tympanic membrane perforation
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will be blinded to the type of barrier received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascia (Active Comparator): Autologous donor substrate
  Interventions: Other: Fascia
- Skye Barrier (Experimental): Amniotic membrane allograft
  Interventions: Other: Skye Barrier

INTERVENTIONS:
Other: Skye Barrier — Substrate derived from amniotic tissue that is FDA-approved for human implantation
  Arms: Skye Barrier
Other: Fascia — Autologous donor substrate. Examples include tragal cartilage, perichondrium, temporalis fascia, and temporoparietal fascia
  Arms: Fascia

SUMMARY:
The trial seeks to provide evidence that the Skye ActiveBarrier provides similar surgical and functional outcomes as fascia when used for tympanoplasties while offering benefits including reduced operative time, better patient satisfaction, and fewer complications.

DETAILED DESCRIPTION:
A prospective randomized controlled trial will be conducted. Eligible patients will be identified, recruited and randomized to receive either repair using the standard fascia graft or repair using the Skye ActiveBarrier. Subjects will undergo a preoperative evaluation followed by TM repair and subsequent regular office visits to assess functional outcomes, complications, and satisfaction. Patients will be blinded to the substrate used for their repair. As there are two different approaches for a tympanoplasty (through the ear canal or incision behind the ear) based on the subject's ear anatomy and location of the perforation, a sham surgery will not be necessary to disguise which graft is received. At follow up visits, photos may be taken of patients' TMs and these photos will be evaluated for healing by an otologist who did not conduct the surgery in a blinded fashion. At the 1 year follow up appointment, subjects will be told which substrate they received and at the study's conclusion subjects will notified about the study's findings.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of a tympanic membrane perforation
2. Patient at PI's clinic

Exclusion Criteria:

1. Presence of cholesteatoma
2. Prior surgery on the same-sided TM or middle ear
3. Ossicular chain abnormalities
4. Congenital deformities involving the middle ear or eustachian tube
5. Refusal to undergo surgery

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Comparable or improved performance of Skye ActiveBarrier | 12-18 months
  Comparable or improved performance will be assessed by combining data from 6 specific measurements: air and bone gap audiogram, word recognition score via audiogram, number of surgical/post-surgical complications, operating time and healing time.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaldo Rivera, M.D., Principal Investigator — University of Missouri-Columbia

IPD SHARING:
Plan to Share IPD: No
The investigators do not intend to share individual participant data to other researchers. Analyzed data will be published in peer-review journal.